CLINICAL TRIAL: NCT06195917
Title: Evaluation of the Safety, Effectiveness and Usability of Robotic-assisted Interventional Percutaneous Transhepatic Puncture: A First-in-human Pilot Study
Brief Title: Robotic-assisted Percutaneous Transhepatic Puncture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Professor, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRob-Zhongda001
Record Dates: First submitted 2023-12-07; First posted 2024-01-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Robotic-assisted Interventional Percutaneous transhepatic puncture
  Interventions: Device: Robotic-assisted Interventional Percutaneous transhepatic puncture

INTERVENTIONS:
Device: Robotic-assisted Interventional Percutaneous transhepatic puncture — Robotic-assisted Interventional Percutaneous transhepatic puncture

SUMMARY:
This is a first-in-man study to investigate the feasibility and safety profile of the newly developed robotic system for percutaneous transhepatic interventional procedures, including biopsy and ablation. Participants who were clinically assessed in need of a liver lesion puncture were included in this study.

DETAILED DESCRIPTION:
In current clinical practice, surgeons mainly use personal experience as a judgment criterion to determine the insertion Angle and trajectory of the needle path. In the process of puncture surgery, surgeons will complete the positioning puncture in three-dimensional space based on the guidance of two-dimensional images and personal judgment. Among them, the lack of three-dimensional sense of space in two-dimensional images may cause inaccurate positioning of the puncture needle in three-dimensional space, and even lead to the deviation of the needle tip approach, resulting in inaccurate biopsy sampling or inaccurate anastomosis in the simulation of thermal field before ablation. In addition, during surgery, changes in the patient's own gravity, breathing movements, posture, or the application of force during needle insertion may cause soft tissue displacement, thereby reducing the accuracy of positioning. In general, in order to ensure the accuracy of puncture, doctors will insert needles repeatedly and perform multiple CT scans on patients, which will lead to low surgical efficiency, increased risk of puncture complications, and increased trauma and pain of patients. In addition, in the puncture operation for liver tumors, if the needle insertion path is not accurate and the needle path is adjusted repeatedly, the risk of the puncture needle carrying out tumor cells will increase, which may cause the metastasis and spread of cancer cells, which is also a big challenge for young doctors. The investigators aim to evaluate the safety, effectiveness and usability of robotic-assisted percutaneous transhepatic puncture in this prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older, with no gender restrictions. (2) clinically assessed and deemed in need of a liver lesion puncture. (3) with a intrahepatic lesion no less than 1 cm in diameter. (4)with liver function of Child-Pugh Class A or B. (5) agree to participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. with severe liver cirrhosis or in a decompensated liver function state within the 3 months prior to screening and who have undergone abdominal paracentesis for the treatment of a large amount of ascites.
2. with severe coagulation disorders during the screening period, characterized by a platelet count < 50×10^9/L, a prolonged PT time > 6s, and an international normalized ratio (INR) > 1.5.
3. classified as NYHA heart function Grade III and IV during the screening period.
4. with severe chronic obstructive pulmonary disease (COPD) or severe asthma during the screening period.
5. with renal insufficiency during the screening period, defined by creatinine (Cr) or blood urea nitrogen (BUN/UREA) levels exceeding two times the upper limit of normal.
6. unable to cooperate with surgical positioning and other requirements for surgery.
7. Pregnant or lactating women of childbearing age and other vulnerable groups.
8. have participated in other interventional clinical trials within the month prior to the commencement of this trial.
9. Other individuals who are deemed unsuitable for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
One-time puncture success rate | one day
  One-time puncture success rate is defined as the rate of one-time of successful percutanoues transhepatic puncture

SECONDARY OUTCOMES:
Number of puncture attempts | one day
  Number of puncture attempts was defined as the total number of punctures until the puncture success
Puncture accuracy | one day
  Puncture accuracy was defined as the Euclidean distance to the pre-defined target
Planning time | one day
  Time from completion of the first CT scan to successful surgical planning of the target lesion
Instrument performance evaluation | one day
  The performance of the system was evaluated by investigators, including system display stability evaluation,evaluation of maneuverability and stability of surgical planning cart, evaluation of operation and stability of central control platform,evaluation of maneuverability and stability of optical tracking vehicle,evaluation of maneuverability and stability of robotic manipulator.
Incidence of adverse events | three days
  Safety of the device will be evaluated by reporting the incidence, severity and frequency of all Adverse Events (AE), related and unrelated to the device treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Lu, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Centre of Interventional Radiology and Vascular Surgery, Department of Radiology, Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No